CLINICAL TRIAL: NCT00228137
Title: A Prospective Randomized Double-Blind Study to Assess the Functional Differences Between the PFC and CKS Knee Prostheses
Brief Title: Randomised Controlled Trial PFC Versus CKS Total Knee Prostheses
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Other Study IDs: HJM25577; FBW STRATEC 96856
Record Dates: First submitted 2005-09-13; First posted 2005-09-28 (Estimated); Last update posted 2007-08-09 (Estimated); Status verified 2007-08

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to compare the functional outcome of two different total knee prostheses in a prospective randomised study.

ELIGIBILITY:
Inclusion Criteria:

All patients on the waiting list for a TKA due to an invalidating gonarthrose as a result of osteo-arthrosis or secondary to a rheumatic disease or a trauma.

Exclusion Criteria:

* patient suffering from juvenile rheumatic disease
* patient suffering hemophilia
* patient on the waiting list for posterior stabilized TKA or hinge joint.
* patient who suffers from a lesion of the ligaments due to surgery
* patient who is legally not capable to make decisions
* patient who suffer from cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Start 2002-11; Study Completion 2012-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Maarten MC de Waal Malefijt, MD, Study Chair — Radboud University Medical Center
Locations (1):
- UMC Radboud, Nijmegen, Netherlands

REFERENCES:
- [Derived] Meijerink HJ, Verdonschot N, van Loon CJ, Hannink G, de Waalmalefijt MC. Similar TKA designs with differences in clinical outcome: a randomized, controlled trial of 77 knees with a mean follow-up of 6 years. Acta Orthop. 2011 Dec;82(6):685-91. doi: 10.3109/17453674.2011.636677. Epub 2011 Nov 9. PMID 22066559